CLINICAL TRIAL: NCT01055834
Title: A Bioequivalence Study of Different Formulations of SEP-190 and Food Effect Study in Japanese Healthy Adult Males
Brief Title: A Bioequivalence and Food Effect Study of SEP-190 in Japanese Healthy Subjects (Study SEP 190-102)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 190-102
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-01

CONDITIONS: Insomnia
Keywords: Insomnia; primary insomnia; insomnia associated with psychiatric or physical disorder(s)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

ARMS (2):
- Eszopiclone 3 mg tablet (Experimental)
  Interventions: Drug: Eszopiclone 3 mg
- Eszopiclone 1 mg tablet (Experimental)
  Interventions: Drug: Eszopiclone 1 mg

INTERVENTIONS:
Drug: Eszopiclone 3 mg — Group A Period I, Group B Period II:
  Eszopiclone 3 mg tablet taken orally (po) with water as a single administration in the morning after fasting >=10 hours.
  Except for the water taken with the drug, participants were not allowed any food/ drink from 10 hours before until 4 hours after administration of drug. Except for the water taken with the study drug, participants were not permitted to drink water from 1 hour before until 1 hour after administration of drug.
  Group B Period III:
  Eszopiclone 3 mg tablet taken po with water as a single administration in the morning 30 minutes after the start of breakfast.
  Except for the food/ drink at breakfast and the water taken with the study drug, participants were not allowed any food or drink from 10 hours before until 4 hours after administration of the drug. Except for the food/ drink at breakfast & the water taken with the study drug, participants were not permitted to drink water from 1 hour before until 1 hour after administration.
  Arms: Eszopiclone 3 mg tablet
Drug: Eszopiclone 1 mg — Group A Period II, Group B Period I:
  Eszopiclone three 1 mg tablets (total: 3 mg) taken orally with water as a single administration in the morning after fasting 10 or more hours.
  Except for the water taken with the study drug, participants were not allowed any food or drink (except water) from 10 hours before until 4 hours after administration of the study drug. Except for the water taken with the study drug, participants were not permitted to drink water from 1 hour before until 1 hour after administration of the study drug.
  Arms: Eszopiclone 1 mg tablet

SUMMARY:
The purpose of this study is to investigate and evaluate the bioequivalence and food effect of SEP 190-102 in Japanese healthy subjects by assessing the pharmacokinetics parameters.

ELIGIBILITY:
Inclusion criteria;

1. Participants who are given a full explanation about the objective and details of this study before starting screening and give written consent based on their free will
2. Japanese healthy male adult volunteers
3. Participants who are between 20 and 54 years of age at the time of obtaining written consent
4. Body Mass Index (BMI) is between 18.5 kg/m2 and 25.0 kg/m2 at the time of screening

Exclusion criteria;

1. Participants with a present illness or history of allergy to drug or food, or seasonal allergy
2. Participants who have a known history of any gastrointestinal surgery (e.g., hepatectomy, nephrotomy, etc.) that may affect pharmacokinetic evaluation
3. Participants who are found to have clinically abnormal findings in medical history, symptoms and clinical findings, vital signs, electrocardiograms, or laboratory parameters of which require medical treatment(s), or impaired organ functions
4. Participants who have a known or suspected history of alcohol or drug abuse, or those who have a positive urine drug screening
5. Participants who are positive for hepatitis B surface antigen (HBs antigen), hepatitis C virus (HCV) antibody, or those who are human immunodeficiency virus (HIV)-positive, or those who are positive for syphilis screen
6. Participants who underwent blood transfusion within 12 weeks prior to, those whose 400 mL or more of whole blood was collected within 12 weeks prior to, or those whose 200 mL or more of whole blood was collected within 4 week prior to study drug administration

Ages: 20 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenya Nakai, Study Director — Japan Clinical Pharmacology, Eisai Co., Ltd.
Locations (1):
- Sumida City, Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Eszopiclone One 3 mg Tab First, Then Three 1mg Tabs: Participants received a single dose of Eszopiclone one 3 mg tablet administered orally with water in the morning after fasting for 10 or more hours in Period I. After a washout period of 5 or more days, participants were crossed over and received a single dose of Eszopiclone three 1 mg tablets with water in the morning after fasting for 10 or more hours in Period II. At least a 5 day period passed before post treatment examinations.
- Group B: Eszopiclone Three 1 mg Tabs First, Then One 3 mg Tab: Participants received a single dose of Eszopiclone three 1 mg tablets administered orally with water in the morning after fasting for 10 or more hours in Period I. After a washout period of 5 or more days, participants were crossed over and received a single dose of Eszopiclone one 3 mg tablet with water in the morning after fasting for 10 or more hours in Period II.
  After Period II there was at least a 5 day washout period. Certain participants from Group B who were treated in Period II in the bioequivalence study proceeded to Period III (food effect study) where they received a single dose of Eszopiclone one 3 mg tablet taken orally with water, 30 minutes after the start of breakfast. At least a 5 day period passed before post treatment examinations.
Period: Treatment Period I
Arm/Group | Group A: Eszopiclone One 3 mg Tab First, Then Three 1mg Tabs | Group B: Eszopiclone Three 1 mg Tabs First, Then One 3 mg Tab
Started | 21 | 21
Completed | 20 | 21
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Treatment Period II
Arm/Group | Group A: Eszopiclone One 3 mg Tab First, Then Three 1mg Tabs | Group B: Eszopiclone Three 1 mg Tabs First, Then One 3 mg Tab
Started | 20 | 21
Completed | 20 | 21
Not Completed | 0 | 0
Period: Treatment Period III
Arm/Group | Group A: Eszopiclone One 3 mg Tab First, Then Three 1mg Tabs | Group B: Eszopiclone Three 1 mg Tabs First, Then One 3 mg Tab
Started | 0 (Participants from Group A did not continue into Period III.) | 14 (14 of 21 participants in Group B who were treated in Period II participated in Period III.)
Completed | 0 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Eszopiclone One 3 mg Tab First, Then Three 1mg Tabs: Participants received Eszopiclone one 3 mg tablets administered orally with water in the morning after fasting for 10 or more hours for 3 days in Period I. After a washout period of 5 or more days, participants were crossed over and received Eszopiclone three 1 mg tablets with water in the morning after fasting for 10 or more hours for 3 days in Period II. At least a 5 day period passed before post treatment examinations.
- Group B: Eszopiclone Three 1 mg Tabs First, Then One 3 mg Tab: Participants received Eszopiclone three 1 mg tablets administered orally with water in the morning after fasting for 10 or more hours for 3 days in Period I. After a washout period of 5 or more days, participants were crossed over and received Eszopiclone one 3 mg tablets with water in the morning after fasting for 10 or more hours for 3 days in Period II.
  After Period II there was at least a 5 day washout period. Certain participants from Group B only proceeded to Period III where they received Eszopiclone one 3 mg tablet taken orally with water, 30 minutes after the start of breakfast for 3 days. At least a 5 day period passed before post treatment examinations.
- Total: Total of all reporting groups
Arm/Group | Group A: Eszopiclone One 3 mg Tab First, Then Three 1mg Tabs | Group B: Eszopiclone Three 1 mg Tabs First, Then One 3 mg Tab | Total
Number analyzed (Participants) | 20 | 21 | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 29.3 (6.0) | 33.0 (9.4) | 31.2 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Parameter (Bioequivalence): Maximal Drug Concentration (Cmax)
Description: Pharmacokinetic parameter: maximal drug concentration (Cmax) was measured in order to confirm bioequivalence. Cmax was measured in nanograms per milliliter (ng/mL). Blood sampling was calculated immediately before administration of the study drug and 24 hours after administration of the study drug (0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12, 24 hours post-dose).
Time Frame: immediately before administration & 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12, 24 hours post-dose
Population: Pharmacokinetic analysis set (bioequivalence set): All participants who completed the study and had their samples analyzed, except for one participant in Group A who discontinued the study in Period 1.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Eszopiclone One 3 mg Tablet: Group A Period I, Group B Period II:
  Eszopiclone one 3 mg tablet administered orally as a single administration with water in the morning after fasting for 10 or more hours.
  Except for the water taken with the study drug, participants were not allowed any food or drink (except water) from 10 hours before until 4 hours after administration of the study drug. Except for the water taken with the study drug, participants were not permitted to drink water from 1 hour before until 1 hour after administration of the study drug.
- Eszopiclone Three 1 mg Tablets: Group A Period II, Group B Period I:
  Eszopiclone three 1 mg tablets administered orally as a single administration with water in the morning after fasting for 10 or more hours.
  Except for the water taken with the study drug, participants were not allowed any food or drink (except water) from 10 hours before until 4 hours after administration of the study drug. Except for the water taken with the study drug, participants were not permitted to drink water from 1 hour before until 1 hour after administration of the study drug.
Arm/Group | Eszopiclone One 3 mg Tablet | Eszopiclone Three 1 mg Tablets
Number analyzed (Participants) | 41 | 41
ng/mL | 40.80 (12.39) | 40.21 (11.72)

2. Primary Outcome: Pharmacokinetic Parameter (Bioequivalence): Area Under the Plasma Concentration- Time Curve From Time 0 to Time 24 Hours (AUC[0-24])
Description: Pharmacokinetic parameter: Area under the plasma concentration- time curve from time 0 (administration of the drug) to time 24 hours was measured in order to confirm bioequivalence. AUC was measured in nanogram hours per milliliter (ng*h/mL). Blood sampling was calculated immediately before administration of the study drug and 24 hours after administration of the study drug (0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12, 24 hours post-dose).
Time Frame: immediately before administration & 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12, 24 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Eszopiclone One 3 mg Tablet | Eszopiclone Three 1 mg Tablets
Number analyzed (Participants) | 41 | 41
ng*h/mL | 212.59 (34.18) | 210.03 (31.77)

3. Primary Outcome: Pharmacokinetic Parameter (Food Effect): Maximal Drug Concentration (Cmax)
Description: Pharmacokinetic parameter: maximal drug concentration (Cmax) was measured in order to investigate the effect of food. Cmax was measured in nanograms per milliliter (ng/mL) and was measured under fasted and fed conditions. Blood sampling was calculated immediately before administration of the study drug and 24 hours after administration of the study drug (0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12, 24 hours post-dose).
Time Frame: immediately before administration & 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12, 24 hours post-dose
Population: Pharmacokinetic analysis set (food effect): 14 participants who completed both Period II and Period III, who had been assigned to move on to Period III when assigned to treatment groups.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Eszopiclone One 3 mg Tablet: Group B Period III:
  After Period II there was at least a 5 day washout period. Certain participants from Group B who were treated in Period II in the bioequivalence study proceeded to Period III (food effect study) where they received a single dose of Eszopiclone one 3 mg tablet taken orally with water, 30 minutes after the start of breakfast. At least a 5 day period passed before post treatment examinations.
  Except for the food and drink at breakfast and the water taken with the study drug, participants were not allowed any food or drink (except water) from 10 hours before until 4 hours after administration of the study drug. Except for the food and drink at breakfast and the water taken with the study drug, participants were not permitted to drink water from 1 hour before until 1 hour after administration of the study drug.
Arm/Group | Eszopiclone One 3 mg Tablet
Number analyzed (Participants) | 14
ng/mL
  Fasted Cmax | 37.59 (8.70)
  Fed Cmax | 26.56 (6.75)

4. Primary Outcome: Pharmacokinetic Parameter (Food Effect): Area Under the Plasma Concentration- Time Curve From Time 0 to Time 24 Hours (AUC[0-24])
Description: Pharmacokinetic parameter: Area under the plasma concentration- time curve from time 0 (administration of the drug) to time 24 hours was measured in order to investigate the effect of food. AUC was measured in nanogram hours per milliliter (ng*h/mL) and was measured under fasted and fed conditions. Blood sampling was calculated immediately before administration of the study drug and 24 hours after administration of the study drug (0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12, 24 hours post-dose).
Time Frame: immediately before administration & 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, 12, 24 hours post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Eszopiclone One 3 mg Tablet
Number analyzed (Participants) | 14
ng*hr/mL
  Fasted AUC [0-24] | 199.17 (38.00)
  Fed AUC [0-24] | 194.53 (29.58)

ADVERSE EVENTS:
Description: Safety Analysis Set (bioequivalence): population treated in Period I except for those subjects with no available safety data.
  Safety analysis set (food effect): is defined as the "safety analysis set (bioequivalence)" except for those subjects with no evaluable safety data in Period III.
Groups:
- Eszopiclone One 3 mg Tablet: Eszopiclone one 3 mg tablets administered orally with water in the morning after fasting for 10 or more hours in either first intervention period (Period I) or second intervention period (Period II).
- Eszopiclone Three 1 mg Tablets: Eszopiclone three 1 mg tablets with water in the morning after fasting for 10 or more hours in either first intervention period (Period I) or second intervention period (Period II).
- Eszopiclone One 3 mg Tablet (Fed): After Period II there was at least a 5 day washout period. Certain participants from Group B who were treated in Period II in the bioequivalence study proceeded to Period III (food effect study) where they received a single dose of Eszopiclone one 3 mg tablet taken orally with water, 30 minutes after the start of breakfast. At least a 5 day period passed before post treatment examinations. Adverse Events were collected under fed conditions.
- Eszopiclone One 3 mg Tablet (Fasted): After Period II there was at least a 5 day washout period. Certain participants from Group B who were treated in Period II in the bioequivalence study proceeded to Period III (food effect study) where they received a single dose of Eszopiclone one 3 mg tablet taken orally with water, 30 minutes after the start of breakfast. At least a 5 day period passed before post treatment examinations. Adverse Events were collected under fasted conditions.
Arm/Group | Eszopiclone One 3 mg Tablet | Eszopiclone Three 1 mg Tablets | Eszopiclone One 3 mg Tablet (Fed) | Eszopiclone One 3 mg Tablet (Fasted)
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/41 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 2/42 | 4/41 | 0/14 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eszopiclone One 3 mg Tablet (N=42) | Eszopiclone Three 1 mg Tablets (N=41) | Eszopiclone One 3 mg Tablet (Fed) (N=14) | Eszopiclone One 3 mg Tablet (Fasted) (N=14)
Dysgeusia (Nervous system disorders) | 1 | 3 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No